CLINICAL TRIAL: NCT02581423
Title: Phase IV Clinical Study of Safety and Tolerability of Oral Xeloda (Capecitabine) in Adjuvant Treatment of Resected Cancer of the Colon
Brief Title: A Study of Capecitabine (Xeloda) in the Adjuvant Treatment of Participants With Resected Colon Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18601
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

ARMS (1):
- Capecitabine (Experimental): Participants will receive capecitabine for up to approximately 6 months.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Participants will receive oral capecitabine, 1250 miligrams per meter-squared (mg/m^2) twice daily, in 3-week treatment cycles for up to 8 cycles. Treatment will be administered for 2 weeks followed by 1 week of rest without medication.
  Other Names: Xeloda

SUMMARY:
This study will evaluate the safety and tolerability of capecitabine (Xeloda) in participants who have undergone surgery for colon cancer. Oral Xeloda will be administered twice daily in 3-week cycles for a total of up to 8 cycles. The anticipated time on study treatment is 24 weeks, and the target sample size is 70 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Curative surgery for Stage III colon cancer, performed 4 to 8 weeks before study entry

Exclusion Criteria:

* Macroscopic or microscopic residual tumor
* Evidence of metastatic disease including tumor cells in ascites
* Previous cytotoxic chemotherapy, radiotherapy, or immunotherapy for colon cancer
* Active cardiovascular disease
* Other malignancy within the last 5 years, other than curatively treated basal cell cancer of the skin or in situ cancer of the cervix
* Malabsorption syndrome or lack of physical integrity of the upper gastrointestinal tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 6 months
Incidence of treatment discontinuation due to AEs | Up to approximately 6 months

SECONDARY OUTCOMES:
Incidence of toxocity-related dose reductions | Up to approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (5):
- Bulgaria (5):
  - Blagoevgrad
  - Rousse
  - Shumen
  - Sofia
  - Veliko Tarnovo